CLINICAL TRIAL: NCT00255593
Title: A Prospective, Randomised, Placebo Controlled, Multicenter Study of the Efficacy and Safety of Rituximab as Induction Therapy Together With Tacrolimus, Mycophenolate Mofetil and Steroids for Patients Undergoing Renal Transplantation
Brief Title: Safety and Efficacy Study of Rituximab in Renal Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Eudra CT: 2005-001231-29
Record Dates: First submitted 2005-11-18; First posted 2005-11-21 (Estimated); Last update posted 2007-11-30 (Estimated); Status verified 2007-10

CONDITIONS: Renal Transplantation
Keywords: Kidney; Transplantation; Immunosuppression; Rituximab
MeSH Terms: interventions — Rituximab

INTERVENTIONS:
Drug: rituximab

SUMMARY:
Current strategies for the medical management of transplant patients are largely focused on the prevention and treatment of T-lymphocyte mediated processes. However there is an increasing evidence to suggest that B-lymphocytes have a role in the otherwise classic T-cell mediated rejection of transplants by there ability to act as antigen presenting cells and T-cell activators. Thus there is a significant medical need for effective therapies targeting B cells of transplant patients.One such potential therapy would be to use rituximab, a monoclonal antibody against B-cells in all renal transplant patients. In the present study the efficacy and safety of prophylactic rituximab is studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or above
* Recipients of first or second renal transplants
* Recipients of kidneys from living or cadaveric donors
* Single organ recipients (kidney only)
* Patients providing written informed consent
* Patients cooperative and able to complete all the assessment procedures

Exclusion Criteria:

* Patients receiving other immunosuppressive therapy within the preceding 28 days
* Recipients of HLA-identical sibling kidneys
* Patients with flow-PRA >50% within 6 months prior to enrolment
* Recent history of malignancy
* Active infection
* Pregnant or lactating females
* Women of childbearing potential not willing to use reliable form of contraception

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2005-11; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of biopsyproven rejection, graft loss or death during the first 6 months following transplanation

SECONDARY OUTCOMES:
Renal function at 6 months
Incidence of infections
Incidence of rituximab-related adverse events
Incidence of malignancies

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar E Tydén, Professor, Study Director — Karolinska Institutet
Locations (1):
- Transplantation Surgery, Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Result] Genberg H, Hansson A, Wernerson A, Wennberg L, Tyden G. Pharmacodynamics of rituximab in kidney allotransplantation. Am J Transplant. 2006 Oct;6(10):2418-28. doi: 10.1111/j.1600-6143.2006.01497.x. Epub 2006 Aug 21. PMID 16925569